CLINICAL TRIAL: NCT06615388
Title: Low Energy Availability and Cardiovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Liverpool Hope University (Other)
Collaborators: Oxford Brookes University (Other)
Responsible Party: Sponsor
Other Study IDs: 328540
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Low Energy Availability; Cardiovascular Diseases
Keywords: low energy availability; Cardiovascular Diseases; Physically active females
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Genetic material (DNA) in cells collected from a buccal cheek smear swab test. Methylation analysis (study of cell function) on the buccal cells will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Physically active females: Physically active females with and with low energy availability

SUMMARY:
Low energy availability (LEA) signifies a condition where the body lacks sufficient energy to support essential physiological functions crucial for maintaining optimal health (1). This energy insufficiency can be exacerbated by the demands of sports and exercise, resulting in negative impacts on various physiological, psychological, and sports performance (11, 8, 2). While LEA is commonly associated with cardiovascular abnormalities, such as early atherosclerosis, endothelial dysfunction, and lower blood pressure, the existing body of research faces limitations, including small sample sizes and primarily exploratory approaches (2). Additionally, despite a growing body of evidence suggesting a strong link between DNA methylation (an epigenetic modification influencing gene expression by tagging specific parts of the DNA code) and cardiovascular disease (9, 6), there has been no prior investigation exploring the interplay between DNA methylation, cardiovascular disease, and LEA. To better understand LEA and its effects on cardiovascular health, it is imperative to address these limitations through further research. Utilising more comprehensive markers of cardiovascular disease and expanding the scope of investigations will contribute to a great understanding of LEA and its implications on cardiovascular health (10).

DETAILED DESCRIPTION:
The team plans to include 126 trained to elite female athletes from local sports clubs near the Liverpool area to participate in the study.

Following ethical approval and informed consent from the participants, data will be collected during a one-time visit at Liverpool Hope University in one of the laboratories in the Health Science building.

Following a single laboratory visit, the following will be collected:

1. Demographic data such as age, sports participation (training, competition duration, frequency etc.) and competitive level.
2. Anthropometric data including height, body mass and DEXA scans.
3. Genetic material (DNA) in cells collected from a buccal cheek smear swab test. Methylation analysis (study of cell function) on the buccal cells will be performed.
4. Venous blood samples to determine hormonal profile. For example, measuring for Cholesterol, Lipids, C-reactive protein (CRP), full blood count , BNP (Natriuretic Peptide), Troponin, Oestrogen, GH (growth hormone), Ferritin, Iron studies, B12 and Folate, urea and electrolytes, Liver Function Tests, Calcium, Magnesium, Luteinising hormone, follicle stimulating hormone and sex hormone binding globulin, Prolactin, Cortisol, Progesterone, Testosterone, Insulin, Insulin-like Growth Factor, Thyroid-stimulating hormone, Thyroxine, Triiodothyronine, Creatine kinase and Vitamin D levels.
5. Cardiovascular assessment to test heart and blood vessel health. For example, blood pressure, the stiffness of their arteries, and the thickness of blood vessel walls. Using assessments such as pulse wave velocity (PWV), Carotid Intima-Media Thickness Test (CIMT), Flow-mediated Dilation (FMD) and electrocardiogram (ECG). Pearson r correlation will be performed between Cardiovascular health and Low energy availability variables.
6. Nutritional assessment via 5-day photographic food diaries, weighed food records along with a short interview to ensure accurate readings.
7. Physical activity assessment with accelerometers for seven days to determine physical activity levels. The accelerometers will be dropped off and picked up after one week by the lead researcher, Mr Liam Pope.
8. Eating behaviour and mood tests using the Eating Disorder Examination Questionnaire (EDE-Q) and the Clinical Impairment Assessment (CIA) (12) to assess their eating behaviours.
9. Low energy availability test via the LEAF-Q (5) and calculation of LEA to check if participants are getting enough energy
10. A questionnaire to assess menstrual cycle health, status, and hormonal contraception use
11. Energy expenditure and resting metabolic rate assessment via indirect calorimetry to measure how much energy their bodies use and how much they burn at rest.

In addition, metabolomic analysis, lipoprotein subclass analysis and methylation analysis on blood cells will be performed.

Machine learning models will also be used to detect novel patterns of lipids/metabolites in the data. Multivariate analysis will be performed before the machine learning models.

Two groups will be formed, comprising one group identified as a high LEA risk group and the other as a low LEA risk group. LEA risk status will be established via the Loukes et al. (1999) equation: Energy availability = (Energy intake (kJ) - Energy expenditure during exercise (kJ))/fat-free mass (kg) (5). Group allocation of participants will be based on the following classification: Low risk of LEA High: EA ≥45 kcal/kg LBM/d and high risk of LEA EA 30 kcal/kg LBM/d (3).

To reduce the variability among the participant results concerning their menstrual cycle characteristics, all 126 selected volunteers will engage in a two-month menstrual cycle monitoring process before the testing for the main research study, following the methodological recommendations for female athlete research (7). This monitoring will occur in participants' homes, utilising menstrual cycle tracking apps and ovulation testing kits that will be sent to them. To track menstrual cycles, volunteers will use a menstrual cycle tracking app to record the first and last day of menstruation for each cycle. Daily ovulation tests will also be conducted using urine to detect the mid-cycle surge in luteinising hormone. The occurrence of the mid-cycle surge in luteinizing hormone will be documented in the app, providing visual confirmation to the researcher. This will also serve as crucial information to identify each participant specific menstrual cycle phases.

To ensure consistent testing, the research team will schedule all participants' tests for the main project during their early luteal phase, specifically in phase three. This phase captures a medium oestrogen concentration while keeping progesterone levels low, confirmed by a positive luteinizing hormone surge captured by the ovulation kit. This strategic choice is made to measure hormone levels within a normal range for health assessment, making it easier to identify any potential hormonal imbalances not due to the typical hormonal fluctuations linked with different phases of the menstrual cycle. This approach ensures precise timing aligned with specific menstrual phases that help minimise the impact of cycle-related variations to enhance the main study's results reliability.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender females
* Aged 18 to 35 to avoid recruiting peri or postmenopausal females
* Trained to elite female athletes based on McKay and colleagues' (2021) criteria for participation classification framework. For example, trained (local-level representation), highly trained (competing at the national level) and elite (competing at the international level).
* Females living in the United Kingdom.

Exclusion Criteria:

* Biological Males
* Females aged over 35
* Sedentary females
* Habitual smokers
* Volunteers with any previous experience with Syncope
* Volunteers with any previous diagnosis of ischaemic heart disease, myopathy or any neuromuscular disorder
* Anticoagulants users
* Pregnant women
* Volunteers on lipid-lowering medication
* Taking hormonal contraception (copper IUDs are acceptable)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The team plans to include 126 trained to elite female athletes from local sports clubs near the Liverpool area to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12-13 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to measure the cardiovascular risk factors associated with LEA in trained to elite female athletes. | 1 year

SECONDARY OUTCOMES:
The secondary outcome is to measure the DNA methylation characteristics of trained to elite-level female athletes? | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Hope University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All participant data will be kept confidential in line with GDPR.

REFERENCES:
- [Background] Wasserfurth P, Palmowski J, Hahn A, Kruger K. Reasons for and Consequences of Low Energy Availability in Female and Male Athletes: Social Environment, Adaptations, and Prevention. Sports Med Open. 2020 Sep 10;6(1):44. doi: 10.1186/s40798-020-00275-6. PMID 32910256
- [Background] Mountjoy M, Sundgot-Borgen J, Burke L, Ackerman KE, Blauwet C, Constantini N, Lebrun C, Lundy B, Melin A, Meyer N, Sherman R, Tenforde AS, Torstveit MK, Budgett R. International Olympic Committee (IOC) Consensus Statement on Relative Energy Deficiency in Sport (RED-S): 2018 Update. Int J Sport Nutr Exerc Metab. 2018 Jul 1;28(4):316-331. doi: 10.1123/ijsnem.2018-0136. Epub 2018 May 17. No abstract available. PMID 29771168
- [Background] Melin AK, Heikura IA, Tenforde A, Mountjoy M. Energy Availability in Athletics: Health, Performance, and Physique. Int J Sport Nutr Exerc Metab. 2019 Mar 1;29(2):152-164. doi: 10.1123/ijsnem.2018-0201. Epub 2019 Feb 26. PMID 30632422
- [Background] McKay AKA, Stellingwerff T, Smith ES, Martin DT, Mujika I, Goosey-Tolfrey VL, Sheppard J, Burke LM. Defining Training and Performance Caliber: A Participant Classification Framework. Int J Sports Physiol Perform. 2022 Feb 1;17(2):317-331. doi: 10.1123/ijspp.2021-0451. Epub 2022 Dec 29. PMID 34965513
- [Background] Loucks AB, Verdun M, Heath EM. Low energy availability, not stress of exercise, alters LH pulsatility in exercising women. J Appl Physiol (1985). 1998 Jan;84(1):37-46. doi: 10.1152/jappl.1998.84.1.37. PMID 9451615
- [Background] Kazmi N, Elliott HR, Burrows K, Tillin T, Hughes AD, Chaturvedi N, Gaunt TR, Relton CL. Associations between high blood pressure and DNA methylation. PLoS One. 2020 Jan 30;15(1):e0227728. doi: 10.1371/journal.pone.0227728. eCollection 2020. PMID 31999706
- [Background] Elliott-Sale KJ, Minahan CL, de Jonge XAKJ, Ackerman KE, Sipila S, Constantini NW, Lebrun CM, Hackney AC. Methodological Considerations for Studies in Sport and Exercise Science with Women as Participants: A Working Guide for Standards of Practice for Research on Women. Sports Med. 2021 May;51(5):843-861. doi: 10.1007/s40279-021-01435-8. Epub 2021 Mar 16. PMID 33725341
- [Background] De Souza MJ, Nattiv A, Joy E, Misra M, Williams NI, Mallinson RJ, Gibbs JC, Olmsted M, Goolsby M, Matheson G; Expert Panel. 2014 Female Athlete Triad Coalition Consensus Statement on Treatment and Return to Play of the Female Athlete Triad: 1st International Conference held in San Francisco, California, May 2012 and 2nd International Conference held in Indianapolis, Indiana, May 2013. Br J Sports Med. 2014 Feb;48(4):289. doi: 10.1136/bjsports-2013-093218. PMID 24463911
- [Background] Chilunga FP, Henneman P, Venema A, Meeks KA, Gonzalez JR, Ruiz-Arenas C, Requena-Mendez A, Beune E, Spranger J, Smeeth L, Bahendeka S, Owusu-Dabo E, Klipstein-Grobusch K, Adeyemo A, Mannens MM, Agyemang C. DNA methylation as the link between migration and the major noncommunicable diseases: the RODAM study. Epigenomics. 2021 May;13(9):653-666. doi: 10.2217/epi-2020-0329. Epub 2021 Apr 23. PMID 33890479
- [Background] Black K, Slater J, Brown RC, Cooke R. Low Energy Availability, Plasma Lipids, and Hormonal Profiles of Recreational Athletes. J Strength Cond Res. 2018 Oct;32(10):2816-2824. doi: 10.1519/JSC.0000000000002540. PMID 29624522
- [Background] Areta JL, Taylor HL, Koehler K. Low energy availability: history, definition and evidence of its endocrine, metabolic and physiological effects in prospective studies in females and males. Eur J Appl Physiol. 2021 Jan;121(1):1-21. doi: 10.1007/s00421-020-04516-0. Epub 2020 Oct 23. PMID 33095376
- See also: THE CLINICAL IMPAIRMENT ASSESSMENT QUESTIONNAIRE (CIA) — https://www.credo-oxford.com/pdfs/CIA_3.0_Instructions_for_users.pdf